CLINICAL TRIAL: NCT01549704
Title: Effect of Adductor-Canal-Blockade on High Pain Responders the 1. or 2. Postoperative Day After Total Knee Arthroplasty
Brief Title: Effect of Adductor-Canal-Blockade on High Pain Responders After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Ulrik Grevstad, Consultant, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-UG-11
Record Dates: First submitted 2012-03-01; First posted 2012-03-09 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Pain After Total Knee Arthroplasty
Keywords: Total knee arthroplasty; Adductor canal blockade (ACB); High pain responders; US-guided nerve block
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm RP (Other): first blockade: ropivacaine 7,5mg/ml 30 ml second blockade: placebo: saline 30 ml
  Interventions: Drug: Ropivacaine; Drug: Saline
- Arm PR (Other): first blockade: placebo: saline 30 ml second blockade: ropivacaine 7,5mg/ml 30 ml
  Interventions: Drug: Ropivacaine; Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Arm RP is receiving 30 ml of ropivacaine 7,5 mg/ml at first blockade (ACB) and after 45 minutes another blockade (ACB) with placebo (saline 30 ml).
  Arm PR is receiving 30 ml of placebo (saline) at first blockade (ACB) and after 45 minutes another blockade (ACB)with ropivacaine.
  Other Names: Naropin
Drug: Saline — please see intervention description for ropivacaine
  Other Names: NaCl, placebo

SUMMARY:
The purpose of this study is to determine whether Adductor-Canal-Blockade (ACB) is superior to placebo when it comes to analgetic efficacy in high pain responders after Total Knee Arthroplasty (TKA). High pain responders are defined as patients reporting VAS > 60 during knee flexion the 1. or 2. day after surgery.

DETAILED DESCRIPTION:
The patients will be included the 1. or 2. day after surgery. All TKA patients will be screened. Those reporting VAS > 60 during active 45 degrees knee flexion will be asked to participate.

Included patients will receive 2xACB (singleshot) first placebo (30ml saline) and then ropivacaine (30ml ropivacaine 7,5mg/ml) or the other way around (randomized). There will be 45 minutes between the two blockades. The blockades will be ultrasound guided.

ELIGIBILITY:
Inclusion Criteria:

* TKA within 48 hours and VAS>60 during active 45 degrees knee flexion despite conventional pain medication.
* Informed consent
* ASA 1-3
* BMI 18-40

Exclusion Criteria:

* Unable to communicate in Danish
* Allergic reactions toward drugs used in the
* Abuse of alcohol/drugs
* Unable to cooperate

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Difference in VAS between ACB and placebo during active 45 degrees knee flexion | 45 minutes

SECONDARY OUTCOMES:
Difference in mean VAS between the groups during active knee flexion | 15, 30, 60, 75 and 90 minutes
Difference in mean VAS between the groups at rest | 15, 30, 60, 75 and 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Grevstad, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Grevstad U, Mathiesen O, Lind T, Dahl JB. Effect of adductor canal block on pain in patients with severe pain after total knee arthroplasty: a randomized study with individual patient analysis. Br J Anaesth. 2014 May;112(5):912-9. doi: 10.1093/bja/aet441. Epub 2014 Jan 8. PMID 24401802